CLINICAL TRIAL: NCT02532530
Title: Peri-operative Monitoring of Regional Cerebral Oxygen Saturation and Onset of Delirium in Cardiac Surgery Patients
Brief Title: Peri-operative Monitoring of Cerebral Oxygenation and the Onset of Delirium in Patients Undergoing Cardiac Surgery
Acronym: ICARUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Principal Investigator, prof. dr. Frank Jans, prof. dr., Hasselt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: ZOLDELIRIUM1
Record Dates: First submitted 2015-08-19; First posted 2015-08-25 (Estimated); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Delirium
Keywords: Aortic valve replacement with or without CABG
MeSH Terms: conditions — Delirium | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Other): Adult patients (age ≥ 70 years) undergoing elective on-pump cardiac surgery (i.e. valve replacement with or without 'Coronary Artery Bypass Graft' (CABG) surgery)
  Interventions: Device: Near-Infrared Spectroscopy (NIRS)

INTERVENTIONS:
Device: Near-Infrared Spectroscopy (NIRS) — Near infrared spectroscopy (NIRS) is a non-invasive technique that uses near infrared light between 700 and 1100nm which penetrates several centimeters through skin and bone structures. Light is absorbed by chromophores. There are multiple chromophores which can be detected in the NIR spectrum such as water, lipids, melanin, myoglobin, oxygenated hemoglobin and deoxygenated hemoglobin. Each chromophore has a specific absorption spectrum. By using different wavelengths, it is possible to differentiate chromophores. The difference between oxygenated hemoglobin and deoxygenated hemoglobin can be calculated using the modified Beer-Lambert law, resulting in a numeric value which is a representation of the regional cerebral oxygen saturation.

SUMMARY:
Delirium is an acute brain syndrome characterized by a disturbance in consciousness accompanied by periods of inattention and changes in cognition. Memory impairment, irrelevant speech and disorientation are commonly observed signs and symptoms. Episodes of delirium have been associated with a prolonged hospital stay, functional and cognitive dysfunction and even an increased mortality. Delirium is a common complication in the postoperative setting where the incidence increases with the risk of surgery. The estimated incidence of postoperative delirium after cardiovascular surgery is remarkable, ranging from 31% up to 51%. Diverse preoperative risk factors have been documented for patients undergoing cardiac surgery: age, pre-existing cognitive dysfunction, a history of alcohol abuse and the severity of illness at admission.

An early diagnosis of postoperative delirium is of great importance to prevent long-term cognitive impairment. For this purpose, a highly specific diagnostic monitoring tool should be implemented during perioperative cardiac surgery care. Near infrared spectroscopy (NIRS) provides information on brain oxygenation by quantifying the regional cerebral oxygen saturation (SctO2) at the microvascular level. Recently, two studies showed that preoperative cerebral tissue oxygenation was lower in the cohort of patients that developed delirium postoperatively. Nevertheless, these studies did not investigate whether the onset of postoperative delirium coincided with a change of postoperative SctO2. A relationship between delirium and reduced cerebral blood flow has already been suggested. As such, the occurrence of a postoperative decrease of SctO2 might have been overlooked thus far. Hence, Investigators want to conduct a prospective, interventional study to determine the relationship between postoperative SctO2 and the onset of delirium after cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age ≥ 70 years) undergoing elective on-pump cardiac surgery (i.e. valve replacement with or without Coronary artery bypass graft surgery (CABG))
* Surgery has to be performed under normothermic conditions
* Ability to perform the confusion assessment method for the intensive care unit (CAM-ICU)
* Patients willing to provide written informed consent

Exclusion Criteria:

* Age < 70 years
* Off-pump cardiac surgery
* Surgery performed under hypothermic conditions
* Duration before extubation > 36 hours
* Patients with insufficient knowledge of the Dutch language
* Patients using antipsychotics
* Patients with a known history of alcohol abuse (consuming two or more units a day)

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 103 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Association between changes in cerebral oxygen saturation and postoperative delirium (preoperative) | pre, intra and postoperative measurement of cerebral oxygen saturation (three days)
  The primary objective is to investigate if the development of delirium after cardiac surgery coincides with changes of the cerebral oxygen saturation.

SECONDARY OUTCOMES:
Cerebral autoregulation performance using a COX index | Intraoperative measurement
  Comparison of the cerebral autoregulation using a COX index (correlation between Mean arterial pressure and SctO2) in patients with and without a stage of delirium.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Jans, prof. dr., Principal Investigator — Ziekenhuis Oost-Limburg
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Belgium

REFERENCES:
- [Derived] Eertmans W, De Deyne C, Genbrugge C, Marcus B, Bouneb S, Beran M, Fret T, Gutermann H, Boer W, Vander Laenen M, Heylen R, Mesotten D, Vanelderen P, Jans F. Association between postoperative delirium and postoperative cerebral oxygen desaturation in older patients after cardiac surgery. Br J Anaesth. 2020 Feb;124(2):146-153. doi: 10.1016/j.bja.2019.09.042. Epub 2019 Dec 18. PMID 31862160